CLINICAL TRIAL: NCT02325336
Title: Effect of Bar-code-assisted Medication Administration on Medication Error Rates: a Controlled Randomized Multicentre Trial
Brief Title: Detection Medication Administration Errors Using Bar-code and RFID Technology (DREAM)
Acronym: DREAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K121202
Record Dates: First submitted 2014-12-19; First posted 2014-12-25 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Medication Administered in Error
Keywords: Medication Errors; nurses; hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bar-code-assisted administration (Experimental): during administration rounds, nurses will use the BCMA system to help preventing administration errors
  Interventions: Device: BCMA (bar-code-assisted medication administration)
- control (No Intervention): during administration rounds, nurses will administer drugs as usual

INTERVENTIONS:
Device: BCMA (bar-code-assisted medication administration) — Implementation of ADIM system (Aide a la Distribution Informatisee des Medicaments) which consists of 2 machines with photographic reconnaissance and readers: one for preparation assistance that can be placed at the pharmacy or in the clinical service and one to assist the administration by the nurse in the clinical service.
  In case of discrepancy with the prescription, there is a visual alert. However, the alert can be override by the nurse if she/he gives a justification.
  Other Names: ADIM preparation; ADIM administration
  Arms: bar-code-assisted administration

SUMMARY:
Serious medication administration errors are common in hospitals. Various interventions were developed to help prevention of such errors such as bar-code technology. Investigators aimed to study the effect of bar-code-assisted medication administration (BCMA) system on the rate of medication errors in two hospitals.

They will conduct a randomized controlled trial in 6 care units of two hospitals in Paris, France. Each unit will be randomized in either the control group or the intervention group using the bar-code system to help drug administration. The observation method will be used to evaluate the error rates in the 2 groups at baseline and when BCMA will be implanted. Nurses of the unit will be randomized to determine who will be observed during the administration rounds.

Considering the results of a passed observational study in 4 units (Berdot, BMC Health Serv Research 2012) and the results of the study by Poon and al. (NEJM 2010), investigators estimated that 5.981 TOE (Total Opportunities for Errors) are needed to detect a relative reduction of 45% of error rate.

DETAILED DESCRIPTION:
The ADIM system (Aide a la Distribution Informatisee des Medicaments) consists of 2 machines with photographic reconnaissance and readers: one for preparation assistance that can be placed at the pharmacy or in the clinical service and one to assist the administration by the nurse in the clinical service.

The system ADIM preparation consists of a working area with 2 reader devices (a RFID reader and a bar code reader) and a touch screen . It allows selection from the list of patients, the patient's prescription for which the preparation will be made. It is linked to the drug data base.

The system ADIM administration is composed of a laptop with touch screen, 2 readers (a RFID reader and a barcode reader) , the elements needed to care and a work plan and drawers containing unit dose drugs for patients for a specific nurse. The nurse scans her/his badge, the patient's wristband and each dose administered and prepared by the pharmacy. If the dose is not prepared by the pharmacy, the nurse takes the dose in the automat cabinet. The nurse scans the drug's barcode or select on the touch screen the drug and the required dose of the drug. In case of discrepancy with the prescription, there is a visual alert. However, the alert can be override by the nurse if she/he gives a justification.

ELIGIBILITY:
Inclusion Criteria:

* Nurses of the 6 care units who have drugs to deliver during medication administration rounds will be included

Exclusion Criteria:

* Nurses who refuse to be observed during medication administration rounds and nurses replacement that did not work usually in the studied units will not be included.

Medication administrations during emergencies (e.g., cardiopulmonary resuscitation) will also be excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Medication administration errors rate | one month after the intervention
  Investigators will use the direct-observation method to measure error rates. Observers will shadow staff nurses while administering drugs to patients, without knowing the physician's medication orders, and will record details about the administration. After completing the observation session, medication administration errors will be assessed, by two senior pharmacists, blinded to the unit allocation, by comparing the observed medication administered to the medication intended for that patient. The rate of medication administration errors will be calculated by dividing the number of errors by the total opportunities for errors (TOE). The TOE is defined as the sum of observed administrations and omitted medications. As wrong-time errors are generally considered less severe, overall error rate will be calculated without this type of error.

SECONDARY OUTCOMES:
type of errors | one month after the intervention
  Each administration error will be classified by the two senior pharmacists according to the type of error using the ASHP classification in 9 categories. Wrong-time error is defined as an administration that is early or late by more than 1 hour.
Severity of error | One month after intervention
  Each error will be classified by a multidisciplinary committee according to the potential harm using the NCCMERP classification.
Satisfaction of nurses | One month after intervention
  Satisfaction with the bar-code system will be assessed using a validated questionnaire. It will be filled anonymously by nurses at the end of the observation period in the unit. Evaluation of administration rounds time will be studied also to evaluate satisfaction with the system.
Relevance of the system | One month after intervention
  Relevance of the system will be assessed by studying the system alerts: false negative rates, rates of modifications in preparation/administration of drugs in case of system alerts, rates of unjustified or wrong alerts. During the observation in the intervention group, number and causes of non-use of the bar-code system will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Sabatier, PharmD, PhD, Study Chair — Hopital Europeen Georges Pompidou